CLINICAL TRIAL: NCT06902272
Title: A Phase 2 Study of Circulating Tumor DNA to Predict Response to Neoadjuvant Treatment and De-escalation Adjuvant Immunotherapy in Early-Stage NSCLC (DNA-PREDICT)
Brief Title: ctDNA to Predict Response to Chemo-Immunotherapy and Detect Minimal Residual Disease in Non-Small Cell Lung Cancer
Acronym: DNA-PREDICT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Richa Dawar, MD, Medical Doctor, Oncology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240140
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ctDNA Monitoring Group (Experimental): Participants in this group will receive ctDNA monitoring in combination with standard of care (SOC) Pembrolizumab, SOC platinum doublet chemotherapy, and SOC surgery for resection of tumor.
  Total participation duration is up to 2.5 years.
  Interventions: Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay; Drug: Pembrolizumab; Drug: Platinum Doublet Chemotherapy

INTERVENTIONS:
Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay — ctDNA will be measured in participants in person via blood samples during Screening/Baseline and at the following intervals during treatment and follow-up:
  * During Neoadjuvant Therapy: Approximately once after four cycles of standard of care Pembrolizumab and platinum doublet therapy.
  * Approximately once two weeks before surgery.
  * Approximately once three weeks after surgery.
  * During Adjuvant Therapy: Approximately once every 12 weeks during standard of care, adjuvant Pembrolizumab therapy.
  * Follow-up Period: Approximately once every three months for up to one year.
Drug: Pembrolizumab — Participants will receive standard of care, neoadjuvant Pembrolizumab therapy intravenously (IV) on Day 1 of each three-week cycle, for up to four cycles prior to standard of care surgery. After surgery, low-risk participants may continue standard of care, adjuvant Pembrolizumab therapy for up to six months; high-risk participants may receive standard of care, adjuvant Pembrolizumab therapy for up to 12 months.
Drug: Platinum Doublet Chemotherapy — Participants will receive neoadjuvant platinum doublet chemotherapy intravenously (IV) per standard of care on Day 1 of each three-week cycle for up to four cycles, prior to standard of care surgery. Possible platinum doublet chemotherapy regimens are Cisplatin/Carboplatin in combination with Pemetrexed or Docetaxel or Gemcitabine. Participants receiving Gemcitabine therapy will be administered Gemcitabine, per standard of care, on Day 8 of each three-week cycle.

SUMMARY:
The purpose of this study is to determine if a blood test called circulating tumor DNA (ctDNA) can be used to predict how well patients will respond to treatment and if there is any cancer left after surgery. The investigators will also study if a drug called pembrolizumab can help prevent the cancer from coming back in patients who are ctDNA-positive or who have evidence of cancer after treatment and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants must be males or females ≥18 years of age on day of signing the informed consent form.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
3. Participants with histologically confirmed Stage IB (≥4 cm), II, or IIIB (N2) NSCLC (as per the 8th American Joint Committee on Cancer (AJCC)) who are considered resectable by a multidisciplinary team and who are going to be treated with neoadjuvant treatment including chemotherapy, immunotherapy, and in some cases radiation before surgery
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
5. Participants must have tumor tissue available for programmed cell death ligand 1 (PD-L1) immunohistochemical (IHC) testing performed by a third-party analyzing lab during the screening period:

   1. Either a formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections, with an associated pathology report, must be submitted for biomarker evaluation prior to randomization. The tumor tissue sample may be fresh or archival if obtained within 6 months prior to enrollment
   2. Tissue must be a core needle biopsy, excisional or incisional biopsy. Fine needle biopsies obtained by endobronchial ultrasound (EBUS) are not considered adequate for biomarker review and randomization. Core needle biopsies obtained by EBUS are acceptable for randomization.

Exclusion Criteria:

1. Presence of locally advanced, unresectable, or metastatic disease. Mediastinal lymph node samples at levels 4 (bilaterally) and 7 are required for clinical staging to assess nodal involvement in participants with mediastinal adenopathy on positron emission tomography-computed tomography scan (PET/CT).
2. Participants with known epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) translocation
3. Previous exposure to anti-cancer therapy, including chemotherapy, radiotherapy or immunotherapy, and previous exposure to immunosuppressive drugs within 3 weeks before neoadjuvant treatment
4. Participants with impaired decision-making capacity .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-06-11 (Estimated); Study Completion 2029-06-11 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA Clearance: Neoadjuvant Phase Measured by Percentage of Participants | Baseline, 3 months
  ctDNA clearance is defined as change from detectable ctDNA at start of neoadjuvant treatment to no detectable ctDNA at the end of neoadjuvant treatment or prior to surgery. The percentage of participants experiencing ctDNA clearance will be reported.
Pathologic Complete Response (pCR) As Measured By Percentage of Participants | Up to 3 months
  Pathologic Complete Response (pCR) is defined as percentage of participants who underwent surgery after neoadjuvant therapy with 0% viable tumor in resected lung and lymph nodes.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 2.5 years
  Recurrence-free survival (RFS) is the elapsed time in months from the date of surgery until the first documented date of local recurrence, distant relapses (recurrence will be assessed by imaging; distant relapses will be assessed by imaging), or death from any cause, whichever is earlier. For alive patients without recurrence/relapse, follow-up time will be censored at the last documented date of disease assessment.
Overall survival (OS) | Up to 2.5 years
  Overall survival (OS)is the elapsed time in months from the date of surgery until the date of death. For alive patients, follow-up time will be censored at the last date known to be alive.
Percentage of Participants Achieving ctDNA Clearance: Adjuvant Phase | Up to 1.5 years
  ctDNA clearance is defined as detectable ctDNA at start of adjuvant treatment to no detectable ctDNA during the post-operative period. The percentage of participants experiencing ctDNA clearance will be reported.
Percentage of Participants With ctDNA Recurrence: Adjuvant Phase | Up to 1.5 years
  ctDNA recurrence is defined as no detectable ctDNA at the start adjuvant treatment initiation to detectable ctDNA during the post-operative period. The percentage of participants with ctDNA recurrence will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Richa Dawar, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No